CLINICAL TRIAL: NCT06382311
Title: A PHASE 1/2, RANDOMIZED, PARTIALLY-BLIND, DOSE-FINDING/DOSE-CONFIRMATION STUDY TO EVALUATE THE SAFETY, REACTOGENICITY AND IMMUNOGENICITY OF THE MRNA-BASED INVESTIGATIONAL PANDEMIC H5 INFLUENZA VACCINE CANDIDATE ADMINISTERED IN HEALTHY YOUNGER AND OLDER ADULTS
Brief Title: A Study to Find and Confirm the Dose and Assess Safety, Reactogenicity and Immune Response of a Vaccine Against Pandemic H5N1 Influenza Virus in Healthy Younger and Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 221824
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Influenza, Human
Keywords: Influenza A virus; Avian influenza; Flu pandemic; Healthy younger adults; Healthy older adults; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner in Phase 1 and Phase 2 Part A.
  Phase 2 Part B: 2 sub-cohorts: Observer-blind and Open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (27):
- Flu mRNA_Ph1_1_YA (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 1 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 1
- Flu mRNA_Ph1_2_YA (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 2 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 2
- Flu mRNA_Ph1_3_YA (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 3 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 3.
- Flu mRNA_Ph1_4_YA (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 4 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 4
- Flu mRNA_Ph1_5_YA (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 5 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 5
- Placebo_Ph1_YA (Placebo Comparator): YA participants receive 2 doses of Placebo during Phase 1, at Day 1 and at Day 22.
  Interventions: Drug: Placebo
- Flu mRNA_Ph1_1_OA (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 1 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 1
- Flu mRNA_Ph1_2_OA (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 2 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 2
- Flu mRNA_Ph1_3_OA (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 3 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 3.
- Flu mRNA_Ph1_4_OA (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 4 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 4
- Flu mRNA_Ph1_5_OA (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 5 during Phase 1, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 5
- Placebo_Ph1_OA (Placebo Comparator): OA Adult participants receive 2 doses of Placebo during Phase 1, at Day 1 and at Day 22.
  Interventions: Drug: Placebo
- Flu mRNA_Ph2_1_YA Part A (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 1 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 1
- Flu mRNA_Ph2_2_YA Part A (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 2 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 2
- Flu mRNA_Ph2_3_YA Part A (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 3 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 3.
- Flu mRNA_Ph2_4_YA Part A (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 4 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 4
- Flu mRNA_Ph2_5_YA Part A (Experimental): YA participants receive 2 doses of Flu Pandemic mRNA_Dose level 5 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 5
- Placebo_Ph2_YA Part A (Placebo Comparator): YA participants receive 2 doses of Placebo during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Drug: Placebo
- Flu mRNA_Ph2_1_OA Part A (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 1 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 1
- Flu mRNA_Ph2_2_OA Part A (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 2 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 2
- Flu mRNA_Ph2_3_OA Part A (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 3 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 3.
- Flu mRNA_Ph2_4_OA Part A (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 4 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_ Dose level 4
- Flu mRNA_Ph2_5_OA Part A (Experimental): OA participants receive 2 doses of Flu Pandemic mRNA_Dose level 5 during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 5
- Placebo_Ph2_OA Part A (Placebo Comparator): OA participants receive 2 doses of Placebo during Phase 2 Part A, at Day 1 and at Day 22.
  Interventions: Drug: Placebo
- Flu mRNA_Ph2 Part B (Experimental): Participants receive 2 dose of Flu Pandemic mRNA dose level 6 in Phase 2 Part B, at Day 1 and at Day 22.
  Interventions: Biological: Flu Pandemic mRNA_Dose level 6
- Influenza Virus Vaccine_Ph2 Part B (Active Comparator): Participants receive 2 doses of influenza virus vaccine administered in Phase 2 Part B, at Day 1 and at Day 22.
  Interventions: Biological: Influenza virus vaccine
- Placebo_Ph2 Part B (Placebo Comparator): Participants receive 2 doses of Placebo during Phase 2 Part B, at Day 1 and at Day 22.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Flu Pandemic mRNA_Dose level 1 — 2 doses of study intervention are administered to participants intramuscularly.
  Arms: Flu mRNA_Ph1_1_OA; Flu mRNA_Ph1_1_YA; Flu mRNA_Ph2_1_OA Part A; Flu mRNA_Ph2_1_YA Part A
Biological: Flu Pandemic mRNA_Dose level 2 — 2 doses of study intervention are administered to participants intramuscularly.
  Arms: Flu mRNA_Ph1_2_OA; Flu mRNA_Ph1_2_YA; Flu mRNA_Ph2_2_OA Part A; Flu mRNA_Ph2_2_YA Part A
Biological: Flu Pandemic mRNA_ Dose level 3. — 2 doses of study intervention are administered to participants intramuscularly.
  Arms: Flu mRNA_Ph1_3_OA; Flu mRNA_Ph1_3_YA; Flu mRNA_Ph2_3_OA Part A; Flu mRNA_Ph2_3_YA Part A
Biological: Flu Pandemic mRNA_ Dose level 4 — 2 doses of study intervention are administered to participants intramuscularly.
  Arms: Flu mRNA_Ph1_4_OA; Flu mRNA_Ph1_4_YA; Flu mRNA_Ph2_4_OA Part A; Flu mRNA_Ph2_4_YA Part A
Biological: Flu Pandemic mRNA_Dose level 5 — 2 doses of study intervention are administered to participants intramuscularly.
  Arms: Flu mRNA_Ph1_5_OA; Flu mRNA_Ph1_5_YA; Flu mRNA_Ph2_5_OA Part A; Flu mRNA_Ph2_5_YA Part A
Biological: Flu Pandemic mRNA_Dose level 6 — 2 dose of study intervention is administered to participants intramuscularly.
  Arms: Flu mRNA_Ph2 Part B
Biological: Influenza virus vaccine — 2 doses of Influenza virus vaccine are administered to participants intramuscularly.
  Arms: Influenza Virus Vaccine_Ph2 Part B
Drug: Placebo — 2 doses of Placebo are administered intramuscularly to participants in Phase 1 and Phase 2 Part A and 2 dose is administered to participants in Phase 2 Part B.
  Arms: Placebo_Ph1_OA; Placebo_Ph1_YA; Placebo_Ph2 Part B; Placebo_Ph2_OA Part A; Placebo_Ph2_YA Part A

SUMMARY:
The aim of this study is to evaluate the safety, reactogenicity and immunogenicity of the Flu Pandemic messenger RNA (mRNA) vaccine (including dose-finding and dose-confirmation) administered in healthy adults 18 to 85 years of age.

DETAILED DESCRIPTION:
Phase 1 (Ph1) of the study aims to evaluate the reactogenicity, safety, and immunogenicity of 5 dose levels of the investigational vaccine, compared with a placebo, in both younger adults (YA) and older adults (OA). Participants will receive two doses, 21 days apart, with safety data collected up to Day 29. The data from this phase will support the safety evaluation of the assessed dose levels and enable further assessment in higher number of participants in Phase 2 Part A.

Phase 2 (Ph2) Part A will assess the immunogenicity, reactogenicity, and safety of the same 5 dose levels evaluated in Phase 1, with the aim of identifying the doses to proceed to Phase 2 Part B.

Phase 2 Part B will descriptively characterize the dose level of the Flu Pandemic mRNA vaccine candidate selected from Phase 2 Part A, comparing it to an influenza vaccine in a 2-dose schedule. It will also assess safety, reactogenicity, and the immune response induced by the influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between and including 18 and 64 yoa (i.e., 64 years + 364 days; YAs) or between and including 65 and 85 yoa (i.e., 85 years + 364 days; OAs) at the time of the first study intervention administration.
* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, return for follow-up visits).
* Body mass index (BMI) more than or equal to (≥)18 kilogram per square meter (kg/m²) and less than or equal to (≤) 35kg/m².
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants or medically stable patients as established by medical history, clinical examination, and screening safety laboratory assessments (Where applicable) Participants with chronic medical conditions with or without specific treatment (e.g., chronic metabolic, cardiac, pulmonary, renal, hepatic, neurologic, and hematologic diseases) are allowed to participate in this study, if considered by the investigator as medically stable. A stable medical condition is defined as disease not requiring change in therapy or hospitalization for worsening disease during 3 months before enrollment.
* Females of nonchildbearing potential may be enrolled in the study.
* Females of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test at Screening Visit (if applicable) and on the day of each study intervention administration, and
  * has agreed to continue adequate contraception for at least 1 month after completion of the last dose of study intervention.

Exclusion Criteria:

Medical conditions

* Where applicable, FDA toxicity grades will be exclusionary.
* Planned administration of an influenza vaccine before Day 43 time point.
* Current or past malignancy, unless completely resolved without clinically significant sequelae (e.g., no evidence of disease following successful treatment of basal cell carcinoma cases are allowed) for >5 years.
* Has any medical disease or psychiatric condition that, in the opinion of the investigator, precludes study participation because it would place the participant at an unacceptable risk of injury, would render them unable to meet the requirements of the protocol, or may interfere with successful completion of the study.
* Has a bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following intramuscular (IM) injections.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection, based on medical history and physical examination (no laboratory testing required). However, in Phase 2, HIV-infected individuals may be enrolled if they have been stable on antiretroviral therapy for the past 6 consecutive months, i.e., their treatment has not been modified, their CD4 cell count is ≥200/mm³ and their viral load has been undetectable (i.e., HIV-RNA <50 copies/mL) (based on medical records, no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s) (including polyethylene glycol, aminoglycoside antibiotics and egg products).
* History of uncontrolled neurological disorders or seizures, including Guillain-Barré syndrome and Bell's palsy, with the exception of febrile seizures during childhood.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* History of or current suspicion of myocarditis or pericarditis (including following administration, of an mRNA vaccine); or idiopathic cardiomyopathy, or presence of any medical condition that increases the risk myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis, eosinophilic granulomatosis with polyangiitis and persistent myocardial infection.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine, or invasive medical device) other than the study intervention(s) during the period beginning 28 days before the dose of study intervention(s) (Day -28 to Day 1), or their planned use during the study period.
* Administration of a vaccine not foreseen by the study protocol in the period starting 28 days before the study intervention administration or planned administration within 21 days after the (last) study intervention administration*.

  *If emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced to 7 days if, necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.
* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

  * Up to 3 months prior to the study intervention administration:
  * For corticosteroids, this will mean prednisone equivalent 20 mg/day. Inhaled, intra-articular and topical corticosteroids are allowed. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study vaccine administration.
  * Up to 3 months prior to study intervention administration: long-acting immune-modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.
* Administration of immunoglobulins and/or any blood products or plasma derivatives within 3 months before study intervention administration through end of study.

Prior/concurrent clinical study experience

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).
* Participated in an A(H5) influenza vaccine study in the past or have a history of A(H5) influenza infection prior to dosing in this study. This includes influenza subtypes A(H5N1), A(H5N8), A(H5N6).

Other exclusion criteria

* Pregnant or lactating female participant.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 1 months after completion of the vaccination series.
* Has a history of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Any study personnel or their immediate dependents, family, or household members.
* Participants with extensive tattoos covering deltoid region on both arms that would preclude the assessment of local reactogenicity.
* Planned move during the study period that will prohibit participating in the study until study end.
* Donation of blood 3 months prior to the study intervention administration and during the study period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 991 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with solicited administration site events [Phase 1 and Phase 2 Part A] | From Day 1 to Day 7
  The assessed solicited administration site events are pain at administration site, redness at administration site, swelling at administration site and lymphadenopathy.
Percentage of participants with solicited administration site events [Phase 1 and Phase 2 Part A] | From Day 22 to Day 28
  The assessed solicited administration site events are pain at administration site, redness at administration site, swelling at administration site and lymphadenopathy.
Percentage of participants with solicited systemic events [Phase 1 and Phase 2 Part A] | From Day 1 to Day 7
  The assessed solicited systemic events are fever, headache, myalgia, arthralgia, fatigue, and chills. Fever is defined as temperature greater than or equal to (>=)38 degrees Celsius (°C)/ 100.4 Fahrenheit (°F) regardless the location of measurement.
Percentage of participants with solicited systemic events [Phase 1 and Phase 2 Part A] | From Day 22 to Day 28
  The assessed solicited systemic events are fever, headache, myalgia, arthralgia, fatigue and chills. Fever is defined as temperature greater than or equal to (>=)38 degrees Celsius (°C)/ 100.4 Fahrenheit (°F) regardless the location of measurement.
Percentage of participants with unsolicited adverse events (AEs) [Phase 1 and Phase 2 Part A] | From Day 1 to Day 21
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs.
Percentage of participants with unsolicited adverse events (AEs) [Phase 1 and Phase 2 Part A] | From Day 22 to Day 42
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs.
Percentage of participants with medically attended adverse events (MAAEs) [Phase 1 and Phase 2 Part A] | From Day 1 to Day 203
  An MAAE is defined as an unsolicited AE for which the participant receives medical attention such as hospitalization, or an emergency room visit, or visit to/by a health care provider.
Percentage of participants with serious adverse events (SAEs) [Phase 1 and Phase 2 Part A] | From Day 1 to Day 203
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, abnormal pregnancy outcomes, is a suspected transmission of any infectious agent via an authorized medicinal product.
Percentage of participants with adverse events of special interest (AESIs) [Phase 1 and Phase 2 Part A] | From Day 1 to Day 203
  Events considered as AESIs are severe hypersensitivity reactions and myocarditis/pericarditis.
Phase 1: Percentage of participants with increase in FDA toxicity grading for hematology and clinical chemistry laboratory parameters from baseline to any level of FDA toxicity grading at Day 8 | Baseline (Day 1), Day 8
Phase 1: Percentage of participants with increase in FDA toxicity grading in hematology and clinical chemistry laboratory parameters from baseline to any level of FDA toxicity grading at Day 29 | Baseline (Day 1), Day 29
Phase 1: Percentage of participants with increase in haematology and clinical chemistry laboratory parameters from normal values at baseline to abnormal values at Day 8 | Baseline (Day 1), Day 8
Phase 1: Percentage of participants with increase in hematology and clinical chemistry laboratory parameters from normal values at baseline to abnormal values at Day 29 | Baseline (Day 1), Day 29
Percentage of participants with anti- hemagglutinin inhibition (HI) titers ≥ 1:40 at Day 43 [Phase 1 and Phase 2 Part A] | At Day 43
Percentage of participants with solicited administration site events [Phase 2 Part B] | From Day 1 to Day 7
  The assessed solicited administration site events are pain at administration site, redness at administration site, swelling at administration site and lymphadenopathy.
Percentage of participants with solicited administration site events [Phase 2 Part B] | From Day 22 to Day 28
  The assessed solicited administration site events are pain at administration site, redness at administration site, swelling at administration site and lymphadenopathy.
Percentage of participants with solicited systemic events [Phase 2 Part B] | From Day 1 to Day 7
  The assessed solicited systemic events are fever, headache, myalgia, arthralgia, fatigue, and chills. Fever is defined as temperature >= 38°C/100.4°F regardless the location of measurement. The preferred location for measuring temperature is axillary.
Percentage of participants with solicited systemic events [Phase 2 Part B] | From Day 22 to Day 28
  The assessed solicited systemic events are fever, headache, myalgia, arthralgia, fatigue, and chills. Fever is defined as temperature >= 38°C/100.4°F regardless the location of measurement. The preferred location for measuring temperature is axillary.
Percentage of participants with unsolicited AEs [Phase 2 Part B] | From Day 1 to Day 21
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs.
Percentage of participants with unsolicited AEs [Phase 2 Part B] | From Day 22 to Day 42
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs.
Percentage of participants with MAAEs [Phase 2 Part B] | From Day 1 to Day 203
  MAAE is defined as an unsolicited AE for which the participant receives medical attention such as hospitalization, or an emergency room visit, or visit to/by a health care provider.
Percentage of participants with SAEs [Phase 2 Part B] | From Day 1 to Day 203
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, abnormal pregnancy outcomes, is a suspected transmission of any infectious agent via an authorized medicinal product.
Percentage of participants with AESIs [Phase 2 Part B] | From Day 1 to Day 203
  Events considered as AESIs are severe hypersensitivity reactions, Aminotransferase (AT) elevation and myocarditis/pericarditis.
Percentage of participants with increase in FDA toxicity grading for clinical chemistry laboratory parameters from baseline to any level of FDA toxicity grading at Day 8 [Phase 2 Part B] | Baseline (Day 1), Day 8
Percentage of participants with increase in FDA toxicity grading for clinical chemistry laboratory parameters from baseline to any level of FDA toxicity grading at Day 29 [Phase 2 Part B] | Baseline (Day 1), Day 29
Percentage of participants with increase in clinical chemistry laboratory parameters from normal values at baseline to abnormal values at Day 8 [Phase 2 Part B] | Baseline (Day 1), Day 8
Percentagev of participants with increase in clinical chemistry laboratory parameters from normal values at baseline to abnormal values at Day 29 [Phase 2 Part B] | Baseline (Day 1), Day 29
Percentage of participants with anti-HI titers ≥ 1:40 at Day 43 [Phase 2 Part B] | At Day 43
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 2 Part B] | At Day 43 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer ≥1:40 in the serum of participants with pre-dose titer below 1:10 or as a ≥4-fold rise in post dose HI titers with pre- dose titer ≥1:10.
GMT Ratio of anti-HI antibody titers [Phase 2 Part B] | At Day 43

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) of HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 1, Day 22, Day 29, Day 43, and Day 203
Geometric mean increase (GMI) of HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 22 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the ratios of the post-vaccination to the pre-vaccination titer.
Geometric mean increase (GMI) of anti-HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 29 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
Geometric mean increase (GMI) of anti-HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 43 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
Geometric mean increase (GMI) of anti-HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 203 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
Percentage of participants with HI antibody Seroconversion rate (SCR) [Phase 1 and Phase 2 Part A] | At Day 22 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer ≥1:40 in the serum of participants with pre-dose titer below 1:10 or as a ≥4-fold rise in post dose HI titers with pre- dose titer ≥1:10.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 29 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer ≥1:40 in the serum of participants with pre-dose titer below 1:10 or as a ≥4-fold rise in post dose HI titers with pre- dose titer ≥1:10.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 43 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer ≥1:40 in the serum of participants with pre-dose titer below 1:10 or as a ≥4-fold rise in post dose HI titers with pre- dose titer ≥1:10.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 1 and Phase 2 Part A] | At Day 203 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer ≥1:40 in the serum of participants with pre-dose titer below 1:10 or as a ≥4-fold rise in post dose HI titers with pre- dose titer ≥1:10.
Percentage of participants with anti-HI antibody titers >= 1:40 [Phase 1 and Phase 2 Part A] | At Day 22, Day 29, and Day 203
Percentage of seropositive participants for the HA antibody titers [Phase 1 and Phase 2 Part A] | At Day 1, Day 22, Day 29, Day 43, and Day 203
  Seropositivity is defined as titers ≥ lower limit of quantification (LLOQ) at the defined timepoints.
GMT of Anti-HI antibody titers [Phase 2 Part B] | At Day 1, Day 22, Day29, Day 43 and Day 203
GMI of anti-HI antibody titers [Phase 2 Part B] | At Day 22 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
GMI of anti-HI antibody titers [Phase 2 Part B] | At Day 29 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
GMI of anti-HI antibody titers [Phase 2 Part B] | At Day 43 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
GMI of anti-HI antibody titers [Phase 2 Part B] | At Day 203 compared to pre-vaccination (Day 1, pre-dosing)
  GMI is defined as the geometric mean of the within participant ratios of the post-vaccination anti-HI antibody titer to the pre-vaccination anti-HI antibody titer.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 2 Part B] | At Day 22 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer >=1:40 in the serum of participants with pre-dose titer below 1:10 or as a ≥4-fold rise in post dose HI titers with pre- dose titer >=1:10.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 2 Part B] | At Day 29 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer >=1:40 in the serum of participants with pre-dose titer below 1:10 or as a >=4-fold rise in post dose HI titers with pre- dose titer >=1:10.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 2 Part B] | At Day 43 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer >=1:40 in the serum of participants with pre-dose titer below 1:10 or as a >=4-fold rise in post dose HI titers with pre- dose titer >=1:10.
Seroconversion rate (SCR) of anti-HI antibody titers [Phase 2 Part B] | At Day 203 compared to pre-vaccination (Day 1, pre-dosing)
  HI seroconversion is defined as a post-dose titer >=1:40 in the serum of participants with pre-dose titer below 1:10 or as a >=4-fold rise in post dose HI titers with pre- dose titer >=1:10.
Percentage of participants with anti-HI antibody >= 1:40 [Phase 2 Part B] | At Day 1, Day 22, Day 29, Day 43 and Day 203
Percentage of participants with seropositivity of anti-HI antibody titers [Phase 2 Part B] | At Day 1, Day 22, Day 29, Day 43 and Day 203
  Seropositivity is defined as titers ≥ LLOQ at the defined timepoints.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Chamblee, Georgia
  - GSK Investigational Site, El Dorado, Kansas
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Edmond, Oklahoma
  - GSK Investigational Site, Yukon, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/